CLINICAL TRIAL: NCT06075797
Title: Feasibility of The PediQUEST Response to Pain Of Children With Neurologic Disability (PQ-ResPOND) Intervention: a Pilot Randomized Controlled Trial (RCT)
Brief Title: The PediQUEST Response to Pain Of Children With Neurologic Disability Pilot Randomized Controlled Trial
Acronym: PQ-ResPOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Boston Children's Hospital (Other); Dana-Farber Cancer Institute (Other); University of Alabama at Birmingham (Other); Deakin University (Other)
Responsible Party: Principal Investigator, Joanne Wolfe, MD, MPH, Physician in Chief, Chair, Department of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023p002305; 1R21NR020433 (NIH)
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy Infantile; Disabilities Multiple; Pain
Keywords: Disabled children; pain; palliative care; electronic patient reported outcomes measures; Severe neurologic impairment
MeSH Terms: conditions — Cerebral Palsy; Pain

STUDY DESIGN:
Intervention Model Description: 2:1 parallel RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PQ-ResPOND (Intervention) (Experimental): Participants in the intervention arm will (i) answer weekly PQ-ResPOND Surveys over 12 weeks, (ii) receive feedback reports (generated by the PediQUEST system to summarize parents answers), and (iii) engage with the pediatric palliative care (PPC) team.
  The interprofessional PPC team will focus on child's recurrent pain and related symptoms using a standardized approach and work on family activation strategies.
  Interventions: Behavioral: PediQUEST ResPOND
- Usual care (Control) (No Intervention): Participants randomized to the control arm will be assigned weekly PQ-ResPOND Surveys up to week 12. Participants in this arm will not have access to the full PediQUEST system, i.e. no reports will be generated. They will not meet the PPC team but can receive regular palliative care consultations following the site's usual referral procedures.
  Children in the usual care arm will receive standard care, which at Boston Children's Hospital usually involves several primary clinicians (primarily neurologists or Complex Care Service attending physicians) and access to psychosocial clinician care throughout the illness course. PPC referrals are typically made at the discretion of the primary clinician, often for decision making reasons and/or closer to end-of-life. If a child presents persistent distress, they will be cared through the usual mechanisms. The rationale for collecting weekly surveys is to minimize reporting bias and may increase adherence and retention.

INTERVENTIONS:
Behavioral: PediQUEST ResPOND — PPC teams will have access to feedback reports and the PQ-ResPOND checklist (standardized framework to diagnosis and treatment of recurrent pain behaviors in children with severe neurologic impairment).
  Integration of the PPC team into care will be achieved through (i) initial consultation (goals: identify treatment goals, and address recurrent pain), and (ii) follow-up: the team will contact or visit the family in response to feedback reports or for treatment monitoring purposes.
  Other Names: Intervention Arm
  Arms: PQ-ResPOND (Intervention)

SUMMARY:
The goal of this pilot randomized controlled trial is to test the feasibility of running a full scale randomized controlled trial that compares the effect of the PQ-ResPOND intervention versus usual care to improve recurrent pain in children, adolescents, and young adults with severe neurologic impairment. The main questions it aims to answer are:

* Is the study feasible and acceptable for participants?
* Does PQ-ResPOND have a potential to be effective?

Participants will:

* answer surveys (their parents will) telling us about the child's pain, symptoms, and use of complementary therapies, and about their own psychological distress and satisfaction with care.
* a group will receive the PQ-ResPOND intervention which consists of:

  * activating parents and providers by using the PediQUEST system, a web platform that administers surveys and generates feedback reports alerting parents and providers about the child's experience, AND
  * responding to child pain or discomfort by incorporating the Response team (members of the hospital's palliative care team) into the child's care to privde a standardized approach to managing recurrent pain.

Researchers will use a comparison (control) group consisting of participants who will answer surveys and receive usual care (no feedback reports or consult with palliative care in this group) to see if a randomized design is feasible.

DETAILED DESCRIPTION:
Background: In the US, tens of thousands of children, adolescents, and young adults (AYA) are estimated to live with severe neurologic impairment (SNI). Over 60% of these children endure uncontrolled and often persistent pain, which frequently goes unrecognized and untreated. The impact extends to their parents who commonly experience unremitting physical and psychological distress. There has been a lack of rigorous studies that focus on interventions to alleviate recurrent pain in children with SNI. This gap might be attributed to the stigmatization of these children, who are often from historically marginalized backgrounds, resulting in a low prioritization in research endeavors. To address this inequity and using the ORBIT Model for intervention development, the investigators have adapted and are refining an intervention previously applied in children with cancer. The PediQUEST Response to Pain Of children with Neurologic Disability (PQ-ResPOND) will respond to child distress by using "reciprocal activation" strategies to overcome normalization-the acceptance among parents and clinicians that symptom distress is an unavoidable outcome of serious illness-and integration of a specialty pediatric palliative care team (PPC). The overall objective of the study is to evaluate the feasibility of running a full-scale RCT that compares the effect of the PediQUEST ResPOND intervention vs. usual care in children and AYA with SNI.

Specific Aims are to 1. assess study's feasibility and acceptability by evaluating recruitment (rates and suitability of screening/tracking), adherence to the intervention (by study participants and interventionists), and retention (dropout rates, reasons, and demographics); and, 2. explore potential for intervention's efficacy by estimating effect sizes and variability of the outcomes proposed for the full-scale RCT (child recurrent pain and symptom burden, and parent outcomes) and assessing intervention's acceptability through semi-structured interviews.

Methods: Researchers will conduct a single site Phase II Pilot 2:1 RCT of PQ-ResPOND (intervention, n=30) vs. usual care (control, n=15) in 45 children ≥1 year-old & AYA with SNI and moderate to severe recurrent pain behaviors. After randomization, participants will answer weekly PQ-ResPOND surveys and monthly outcome surveys over 12 weeks via the PQ App, and a semi-structured exit interview. Intervention: participants assigned to this arm will receive the PQ-ResPOND intervention which combines (i) parent-mediated activation through weekly collection and feedback to parents and clinicians, via our PQ App, of parent reported child pain (Non-Communicating Children's Pain Checklist-Revised scale (NCCPC-R)) and other symptoms (PediQUEST-Memorial Symptom Assessment Scale adapted for children with SNI), with (ii) PPC team-mediated activation of primary clinicians and parents: through PPC consultation, and (iii) PPC team activation through training in a standardized approach to recurrent pain using the PQ-ResPOND Checklist (adapted by the study's interprofessional expert panel). Usual care: participants in this arm will continue receiving care as usual.

Outcomes: Investigators will use quantitative and qualitative outcomes to study feasibility and acceptability including recruitment and retention rates, intermittent attrition, adherence to intervention delivery by clinicians, and participant and clinician's acceptability of the intervention. To preliminarily estimate effect sizes and variability, the corresponding scores for child's pain and symptom burden, and parent distress and activation measures will be estimated.

Analysis: For feasibility and acceptability quantitative outcomes investigators will use descriptive statistics. Demographics and reasons for attrition will be reported to explore potential for selection bias. A focused thematic analysis will be used to analyze qualitative variables. To estimate effect sizes and variability of trial outcomes, mixed linear regression models will be estimated. A predefined set of progression criteria are in place.

Discussion: Results will inform whether a full-scale Phase III RCT is warranted, and will help with study design and sample size calculation, development of a manual of procedures and fidelity monitoring strategies.

ELIGIBILITY:
Inclusion Criteria:

* Parent-child dyads will be included based on the following criteria:

Child participants will be selected from the base population of patients who are:

* ≥ 1 year old,
* receiving routine (ongoing) care at Boston Children's Hospital, AND
* followed by the Neurology, Cerebral Palsy or Complex Care services.

All patients from the base population will be screened to include any patient who:

* has severe neurological impairment, defined as:

  * a Central Nervous System disorder resulting in motor and cognitive impairment and an inability to communicate either verbally or through sign language, AND
  * has complete caregiver dependency for activities of daily living AND
* date of diagnosis of SNI is ≥ 4 months prior to the date of screening

Exclusion Criteria:

* Parent-child dyads will be excluded if any of the following apply:

  * the child,

    * is already followed by the palliative care team, OR
    * is not expected to survive at least 2 months after enrollment; OR
    * does not have "moderate to severe recurrent pain", as measured through the baseline Child Pain Survey (PPP). Specifically, we will exclude participants whose:
* "Good days" AND "Difficult days" PPP scores are <14, AND
* "Most troublesome pain" PPP score is <30, AND
* Number of "difficult days" are <8 in past month, AND
* Number of days with "most troublesome pain" are <4 in past month; OR • both parents,

  * do not have legal guardianship, OR
  * are unable to read, write, and speak English OR Spanish
  * are unable to understand and complete surveys.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 16 months
  Proportion of contacted potential participants meeting initial inclusion criteria who consent to participate
Recruitment/month | 16 months
  Number of participants recruited per month
Randomization rate | 16 months
  Proportion of enrolled participants who meet randomization criteria (moderate to severe pain)
Suitability of screening/tracking | 16 months
  Qualitative outcome: As reported by research staff and site investigators involved in patient validation
Sample diversity | 16 months
  Proportion of enrolled participants by race/ ethnicity
Refusal reasons | 16 months
  Qualitative: Description of reasons for refusal mentioned in the consent conversation or non-participation survey
Dropout rate | 16 months
  Proportion of enrolled participants who dropout from the study
Demographics of dropouts | 16 months
  Proportion of dropout participants by race/ ethnicity
Dropout reasons | 16 months
  Description of dropout reasons referred by participants during exit interview or dropout conversation
Intermittent attrition | 16 months
  Surveys' response rates and distribution of non-responses will be used to determine participant's adherence with study data collection procedures
Adherence with answering surveys | 16 months
  Qualitative: Parent perspectives on survey frequency, length, relevance, and burden
Feasibility of intervention delivery | 16 months
  Qualitative: Using information from the PQ system, medical records, and exit interviews we will assess how feasible it is to deliver the different intervention components.
Participant's acceptability of the intervention | At week 12
  Satisfaction with the intervention measured through a numerical 0-10 rating score
Likelihood that participants would recommend study to others | At week 12
  Agreement with recommending the study to others using a numeric 0-10 rating score
Participant's acceptability of intervention (qualitative) | At week 12
  Qualitative: We will explore participant's views on the intervention during exit interviews
Clinician's acceptability of intervention (qualitative) | 16 months
  Qualitative: Clinicians views on the intervention will be explored during semi-structured clinician interviews (these will be conducted every 6 months with a subset of clinicians)
Participant's overall satisfaction with the study | At study exit
  We will analyze participant's overall satisfaction with the study on a 0 to 10 numeric scale

SECONDARY OUTCOMES:
Child pain | 12 weeks
  This is the proposed primary outcome for future Phase III trial. All secondary outcomes will be used to preliminarily estimate effect sizes and help with sample size calculations. We will present estimates of effect, variability, and intraclass correlation coefficients with their 95% Confidence Intervals (95%CI).
  Difference between intervention and control arms of the average Pediatric Pain Profile (PPP) most difficult day of last week scores over 12 weeks, measured monthly, as reported by the parent for all enrolled children. Score range: 0-60, higher scores indicate more pain. Cut off point for pain: 14 (>14 indicates pain)
Child symptom burden | 12 weeks
  Difference between intervention and control arms of the average (PediQUEST ResPOND Memorial Symptom Assessment Scale, PQ-ResPOND MSAS) total scores over 12 weeks, as reported weekly by the parent. PQ-ResPOND MSAS total scores are calculated as the average of the 21 individual symptom scores. Individual symptom scores are calculated as the average of the three symptom questions. Individual symptom scores and total scores range from 0-100, 100 indicates higher symptom burden.
Parent Anxiety | 12 weeks
  Difference between trial arms of the average Spielberger's-State Anxiety Inventory-State scores over 12 weeks, measured monthly. Scores range from 20 to 80, with higher scores correlating with greater anxiety.
Parent Depression | 12 weeks
  Difference between trial arms of the mean Center for Epidemiologic Studies Short Depression Scale (CES-D-10) scores over 12 weeks. Scores range from 0 to 30 (Score of 10 or higher indicates the presence of significant depressive symptoms).
Parent Pain-related Stress | 12 weeks
  Difference between trial arms of the mean pain-related stress scores measured with an adapted version of the stress-portion of the Response to Stress Questionnaire-Pain, measured monthly. The tool assesses 12 potential stress sources. Scores range from 1-4 (higher means more stress). Symptom-related stress score calculated as the sum of the 12 item scores.
Parent overall health quality | 12 weeks
  Difference between trial arms of the mean overall health quality score measured monthly with one item of the Short Form (12) Health Survey (SF-12). Uses a 5 point Likert type scale and is scored 0-100, where 100 is excellent overall health.
Parent sleep quality - total sleep time | 12 weeks
  Parent sleep quality will be measured with an adapted version of the Consensus Sleep Diary. Difference between trial arms of the mean overall score of the weekly average total sleep time (in hours), measured monthly. More hours of sleep is better.
Parent sleep quality - refreshing sleep | 12 weeks
  Measured with an adapted version of the Consensus Sleep Diary. Difference between trial arms of the mean overall weekly score of the refreshing sleep item, measured monthly. Response options 1 to 5, where 5 is extremely refreshing.
Use of Complementary Therapies | 12 weeks
  Difference between trial arms of the No. of complementary therapies used measured monthly with the Use of Complementary therapies checklist (developed ad hoc). Continuous variable, where higher numbers indicates more use of complementary therapies.
Parent Coping - Active coping | 12 weeks
  Difference between trial arms of the mean overall active coping score measured monthly with the Short version of the Coping Orientation to Problems Experienced Inventory (Brief COPE).
  Scores on each scale (or item) range from 2 to 8, with higher scores indicating greater use of that strategy.
Parent Coping - Planning | 12 weeks
  Difference between trial arms of the mean planning coping score measured monthly with the Short version of the Coping Orientation to Problems Experienced Inventory (Brief COPE). Scores on each scale (or item) range from 2 to 8, with higher scores indicating greater use of that strategy.
Parent Coping - Instrumental support | 12 weeks
  Difference between trial arms of the mean instrumental support coping score measured monthly with the Short version of the Coping Orientation to Problems Experienced Inventory (Brief COPE). Scores on each scale (or item) range from 2 to 8, with higher scores indicating greater use of that strategy.
Parent Coping - Acceptance | 12 weeks
  Difference between trial arms of the mean acceptance coping score measured monthly with the Short version of the Coping Orientation to Problems Experienced Inventory (Brief COPE).
  Scores on each scale (or item) range from 2 to 8, with higher scores indicating greater use of that strategy.
Parent Coping - Self-blame | 12 weeks
  Difference between trial arms of the mean self-blame coping score measured monthly with the Short version of the Coping Orientation to Problems Experienced Inventory (Brief COPE). Scores on each scale (or item) range from 2 to 8, with higher scores indicating greater use of that strategy.

OTHER OUTCOMES:
Progression criteria: Recruitment rate | 16 months
  To decide whether to progress or not to a Phase III trial, we will analyze a subset of primary outcomes using a red, amber, green (RAG) approach for each criteria. For recruitment rate we will proceed with RCT (Go) if the indicator is ≥60%, Amend (Proceed with changes) if indicator is between 50% and 59%, and Stop (will not proceed to RCT unless changes are possible) if indicator is <50%.
Progression criteria: Recruitment/month | 16 months
  For recruitment/month we will proceed with RCT (Go) if the indicator is ≥4, Amend (Proceed with changes) if indicator is between 3 and 4 and Stop (will not proceed to RCT unless changes are possible) if indicator is <3 patients/month.
Progression criteria: Retention rate | 16 months
  For retention rate we will proceed with RCT (Go) if the indicator is ≥80%, Amend (Proceed with changes) if indicator is between 70% and 79% and Stop (will not proceed to RCT unless changes are possible) if indicator is <70%.
Progression criteria: Feasibility of intervention delivery | 16 months
  For feasibility of intervention delivery, a qualitative indicator, we will proceed with RCT (Go) if the indicator is judged as strongly feasible, Amend (Proceed with changes) if indicator is judged as feasible, and Stop (will not proceed to RCT unless changes are possible) if indicator is judged as possibly feasible.
Progression criteria: Participant's acceptability of intervention | 16 months
  For participant's acceptability of intervention, a qualitative indicator, we will proceed with RCT (Go) if the indicator is judged (by participants) as strongly acceptable, Amend (Proceed with changes) if indicator is judged (by participants) as acceptable, and Stop (will not proceed to RCT unless changes are possible) if indicator is judged (by participants) as fairly acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Wolfe, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (3):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Deakin University, Burwood, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No